# INFORMATIE VOOR DEELNEMERS AAN MEDISCH-WETENSCHAPPELIJK ONDERZOEK Informatie voor: patiënten na een resectie van een cutaan melanoom

# ONDERZOEK NAAR DE EFFECTEN VAN VEZELRIJKE GEDROOGDE WITLOFWORTEL OP HET DARM MICROBIOOM BIJ OPERATIEF BEHANDELDE MELANOOM PATIËNTEN

Officiële titel van het onderzoek:

Het meten van de effecten van vezelrijke gedroogde witlofwortel op het darm microbioom van patiënten met een gemiddeld tot hoog risico geclassificeerd cutaan melanoom: een exploratieve studie

Officiële Engelse titel van het onderzoek:

Measuring effects of high-fiber dried chicory root on the gut microbiota of patients with intermediate to high-risk cutaneous melanoma: an explorative study

Geachte heer/mevrouw,

Met deze informatiebrief willen we u vragen of u wilt meedoen aan medisch-wetenschappelijk onderzoek speciaal gericht op patiënten na recente verwijdering van een melanoom op de huid. Dit onderzoek richt zich op het toevoegen van vezelrijke gedroogde witlofwortel aan de dagelijkse voeding. Door het toevoegen van voedingsvezels aan de dagelijkse voeding kunnen korte-keten vetzuren door specifieke bacteriën in de dikke darm geproduceerd worden. In eerdere onderzoeken is aangetoond dat er een positieve relatie is tussen korte-keten vetzuren en de gezondheid van de darmen. Deze stofjes dragen bij aan het ondersteunen en onderhouden van een gezonde darmwand.

De informatie in deze brief kunt u rustig doorlezen en naderhand bedenken of u mee wilt doen. Wanneer u mee wilt doen, neem dan contact op de coördinerend onderzoeker. De contactgegevens kunt u vinden in **bijlage A**. Na akkoord zal de onderzoeker een afspraak met u maken waarbij het toestemmingsformulier getekend kan worden. Het toestemmingsformulier vindt u aan het einde van deze brief, bij **bijlage D**. Meedoen is vrijwillig.

## Stel uw vragen

U kunt uw beslissing nemen met de informatie die u in deze informatiebrief vindt. We raden u aan om vragen te stellen aan de onderzoeker die u deze informatie geeft. Verder, is het goed om over dit onderzoek te praten met uw partner, familie of vrienden.

Daarnaast kunt u informatie lezen over overzoek in het algemeen op www.rijksoverheid.nl/mensenonderzoek.

# 1. Algemene informatie

Dit onderzoek is opgezet binnen het UMCG. De uitvoering van het onderzoek vindt plaats binnen het UMCG en wordt gedaan door onderzoekers met kennis over het huidmelanoom, voeding, darmbacteriën en darmgezondheid.

Deelnemers aan een medisch-wetenschappelijk onderzoek worden vaak proefpersonen genoemd. Zowel patiënten als mensen die gezond zijn, kunnen proefpersoon zijn. Voor dit onderzoek zijn ongeveer 20 proefpersonen nodig. De medisch-ethische toetsingscommissie UMC Groningen heeft dit onderzoek goedgekeurd.

## 2. Doel van het onderzoek

In deze studie willen we onderzoeken of het dagelijks gebruik van vezelrijke gedroogde witlofwortel effect heeft op de korte-keten vetzuur productie door specifieke darmbacteriën. Ten tweede willen we weten of het product goed verdragen wordt en de samenstelling van de darmbacteriën bij recent geopereerde melanoom patiënten kan veranderen.

# 3. Achtergrondinformatie

Het is bekend dat er verschillende factoren van invloed kunnen zijn op het terugkeren van het melanoom. Dit terugkeren kan zowel lokaal plaatsvinden of door uitzaaiing via de bloedbaan. Voorbeelden van deze factoren zijn: de dikte van het melanoom en uitzaaiingen in de lymfeklieren. We weten dat bij de behandeling van het melanoom een goed afweersysteem belangrijk is. Een van de factoren die mogelijk belangrijk kan zijn voor de functie van het afweersysteem is de samenstelling van uw darmbacteriën.

Welke bacteriën er in uw darmen leven hangt samen met bepaalde voedingspatronen. Het mediterrane dieet is misschien wel een bekend voorbeeld van zo'n voedingspatroon. Ondanks aangetoonde relaties met het mediterrane dieet, de samenstelling van bacteriën in de darmen en het effect op immuuntherapie bij patiënten met een melanoom, weten we niet welk onderdeel van dit type voedingspatroon het effect veroorzaakt. We weten wel dat het mediterrane dieet bekend staat als een vezelrijk dieet.

Door het toevoegen van voedingsvezels aan de dagelijkse voeding kunnen korte-keten vetzuren door specifieke bacteriën in de dikke darm geproduceerd worden. Om het effect van vezelinname op de vorming van korte-keten vetzuren en de samenstelling van uw darmbacteriën te kunnen bestuderen, gebruiken wij gedroogde witlofwortel in dit onderzoek. Deze gedroogde witlofwortel bevat van nature een hoog gehalte aan voedingsvezels. Dit voedingsproduct zal naast uw reguliere voeding gebruikt worden en dient niet als alternatief voor een gebalanceerde maaltijd.

U gaat het voedingsproduct WholeFiber™ (WholeFiber Holding BV, Espel, Nederland) gebruiken. Dit product is commercieel verkrijgbaar op de Nederlandse markt. De dosis zal 20 g/dag zijn, wat overeenkomt met 17 g voedingsvezels per dag. In de eerste week zal de dosis 10 g/dag zijn, ter gewenning aan het product. Naast voedingsvezels bevat het een laag gehalte aan eiwitten (5%), vet (<1%), mono- en disachariden (3%), organische zuren (2%) en mineralen (2%).

# 4. Verloop van de onderzoeksperiode

De totale onderzoeksperiode bedraagt 6 weken, waarin u gedroogde witlofwortel zult gebruiken naast uw reguliere voeding. Binnen de periode van 6 weken wordt u 3 keer gevraagd worden om naar het UMCG te komen voor onderzoeken en metingen. Deze zijn in detail uitgelegd in 'onderzoeken en metingen'.

## Bent u geschikt om mee te doen?

We willen eerst weten of u geschikt bent om mee te doen. Daarom doet de onderzoeker een aantal onderzoeken:

- Medische geschiedenis uitvragen
- Het bepalen van uw melanoomstatus
- Het bepalen van uw medicatie gebruik

### Het gebruik van het vezel product

U gaat gedurende 6 weken een voedingsvezel product gebruiken. Het onderzoeksmiddel krijgt u mee in zakjes met een dosering van 10 gram. Dit wordt tweemaal daags ingenomen, wat neerkomt op een dagelijkse dosis van 20 gram. In de eerste week van het onderzoek zult u één zakje per dag innemen Het product is te gebruiken naast uw reguliere voeding. U kunt kiezen hoe u het onderzoeksmiddel consumeert, dit kan zonder toevoegingen, door het over de maaltijd heen te strooien of door het in de maaltijd te verwerken. U zult over de manier van consumptie advies krijgen tijdens het eerste onderzoek bezoek.

#### Onderzoeken en metingen

Voor het onderzoek is het nodig dat u in totaal vier keer een afspraak heeft met de onderzoekers, drie van deze afspraken zullen plaatsvinden in het UMCG en het eerste gesprek kan eventueel telefonisch plaatsvinden. Een bezoek duurt gemiddeld 1 uur.

We doen de volgende onderzoeken:

- Lichamelijk onderzoek.
  - De onderzoeker meet uw lengte, gewicht en bloeddruk.
- Onderzoek van uw bloed.

Daarvoor neemt de onderzoeker per keer 1 buisjes bloed af. Wij nemen 3 keer bloed af gedurende de onderzoeksperiode, in totaal is dat 3 buisjes of 30 ml.

Met het bloedonderzoek testen we deze zaken:

- o Eventuele veranderingen in ontstekingswaarden
- o Immuun cel populatie
- Onderzoek van uw ontlasting.

Daarvoor verzamelt u thuis uw ontlasting met behulp van het ontlasting verzamelpakket, wat u ontvangt van de onderzoeker. Het verzamelen van ontlasting kunt u 1-3 dagen voordat de afspraak met de onderzoeker plaatsvindt doen. U neemt de ontlasting mee naar de onderzoek afspraak in de daarvoor bestemde koeltas uit het ontlasting verzamelpakket.

Met het ontlasting onderzoek testen we deze zaken:

- o De samenstelling van de bacteriën in uw darmen
- De productie van korte-keten vetzuren
- o Eventuele veranderingen in ontstekingswaarden
- U vult vragenlijsten in.

De vragen gaan over uw dieet voorafgaand aan de interventie, voedingstoestand, gesteldheid van de darmen en eventuele bijwerkingen die u ervaart.

In **bijlage B** staat welke metingen we doen bij ieder bezoek. Hier staat ook vermeld welke vragenlijsten ingevuld moeten worden voor het bezoek.

## 5. Overeenkomsten met de onderzoekers

We willen graag dat het onderzoek goed verloopt. Daarom maken we graag de volgende afspraken met u:

- U neemt het product in op de manier die de onderzoeker u heeft uitgelegd.
- U geeft aan wanneer u meedoet aan een ander medisch-wetenschappelijk onderzoek.
- U komt iedere afspraak na.

Graag contact opnemen met de onderzoeker in de volgende situaties:

- o U wilt andere medicijnen gaan gebruiken. Ook als dit homeopathische middelen, natuurgeneesmiddelen, vitaminen of geneesmiddelen van de drogist zijn.
- o U wordt in een ziekenhuis opgenomen of behandeld.
- o U krijgt plotseling problemen met uw gezondheid.
- o U wilt niet meer meedoen met het onderzoek.
- o Uw telefoonnummer, adres of e-mailadres veranderd.

# 6. Bijwerkingen, nadelige effecten of ongemakken

Het product bevat een grote hoeveelheid voedingsvezels. Onderzoek deelnemers die normaal gesproken geen vezelrijk dieet volgen, kunnen darmklachten ervaren (bijvoorbeeld een opgeblazen gevoel, winderigheid, diarree, constipatie of krampen) wanneer zij het product consumeren. Deze ongemakken zijn naar verwachting minimaal en mogen in de eerste dagen van gebruik niet langer dan een paar uur duren. In de voorgaande klinische onderzoeken rapporteerden de deelnemers tijdens geen van de vele studiebezoeken enige ernstige bijwerkingen.

Mocht u veel last van de darmen ondervinden waarbij de last ondragelijk is, zal u aangeboden worden om eerst een periode te stoppen met de interventie totdat de klachten niet meer aanwezig zijn. Na deze periode zal u de optie gegeven worden om verder te gaan in de studie met een lagere dosering. Wanneer er toch onverwachte bijwerkingen optreden neem dan contact op met het onderzoeksteam, zie hiervoor de namen en het telefoonnummer onder aan deze brief.

## 7. Voordelen en nadelen van het meedoen aan dit onderzoek

Het vezel product kan de algemene gezondheid van uw darm microbioom verbeteren, maar zeker is dat niet.

Meedoen aan het onderzoek kan deze nadelen of gevolgen hebben:

- U kunt last krijgen van de ongemakken van het vezel product.
- U kunt last hebben van de metingen tijdens het onderzoek.
- Meedoen aan het onderzoek kost u extra tijd.
- Het houden aan de afspraken die horen bij het onderzoek.

## Wilt u niet meedoen?

Geen probleem. U beslist zelf of u deelneemt aan het onderzoek. Uw keuze wordt volledig gerespecteerd en heeft geen invloed op uw verdere behandelingstraject.

# 8. Beëindiging van het onderzoek

De onderzoeker laat het u weten als er nieuwe informatie over het onderzoek komt die belangrijk voor u is. De onderzoeker vraagt u op basis van deze informatie of u wilt blijven meedoen.

In deze situaties stopt voor u het onderzoek:

- Alle onderzoeken volgens het schema (bijlage B) zijn voorbij.
- U wilt zelf stoppen met het onderzoek. Dat mag op ieder moment. Meld dit dan meteen bij de onderzoeker. U bent niet verplicht te vertellen waarom u wilt stoppen.
- De onderzoeker vindt het beter voor u om te stoppen.
- Een van de volgende instanties besluit dat het onderzoek moet stoppen:
  - o Het UMCG
  - o De overheid
  - o De medisch-ethische commissie die het onderzoek beoordeelt

Wanneer u besluit te stoppen met het onderzoek zullen de onderzoekers de verzamelde gegevens en het lichaamsmateriaal (bloed en feces) gebruiken die tot het moment van stoppen zijn verzameld. Als u wilt, kan verzameld lichaamsmateriaal worden vernietigd. Geef dit door aan de onderzoeker. Het gehele onderzoek is afgelopen als alle deelnemers klaar zijn met de onderzoeken volgens het onderzoek schema (bijlage B).

## 9. Na het onderzoek

Het duurt ongeveer één jaar voordat dit onderzoek klaar is. Na uw deelname laat de onderzoeker u weten wat de belangrijkste uitkomsten zijn van het onderzoek. Meldt het aan de onderzoeker wanneer u niet geïnteresseerd bent in de uitkomsten, dan wordt u daarover niet benaderd.

# 10. Opslag en verwerking van gegevens en lichaamsmateriaal

Wanneer u meedoet met het onderzoek, dan geeft u ook toestemming om uw gegevens en lichaamsmateriaal te verzamelen, gebruiken en bewaren.

De volgende gegevens zullen gebruikt en bewaard worden:

- Uw naam
- Uw geslacht
- Uw adres
- Uw geboortedatum
- · Gegevens over uw gezondheid
- Gegevens die we tijdens het onderzoek verzamelen

De volgende lichaamsmaterialen zullen gebruikt en bewaard worden:

- Bloed buisjes die we tijdens het onderzoek verzamelen
- Feces buisjes die we tijdens het onderzoek verzamelen

We verzamelen, gebruiken en bewaren uw gegevens en uw lichaamsmateriaal om de vragen van dit onderzoek te kunnen beantwoorden, en om de resultaten te kunnen publiceren. Om uw privacy te beschermen geven wij uw gegevens en uw lichaamsmateriaal een code. Op al uw gegevens en lichaamsmateriaal zetten we alleen deze code. De sleutel van de code bewaren we in een beveiligde map in het UMCG. Als we uw gegevens en lichaamsmateriaal verwerken, gebruiken we steeds alleen die code. Ook in rapporten en publicaties over het onderzoek kan niemand terughalen dat het over u ging.

Sommige personen kunnen wel uw naam en andere persoonlijke gegevens zonder code inzien. Dit kunnen gegevens zijn die speciaal voor dit onderzoek zijn verzameld, maar ook gegevens uit uw medisch dossier. Dit zijn mensen die controleren of de onderzoekers het onderzoek goed en betrouwbaar uitvoeren.

Deze personen kunnen bij uw gegevens komen:

- Leden van de commissie die de veiligheid van het onderzoek in de gaten houdt.
- Nationale en internationale toezichthoudende autoriteiten.

Deze personen houden uw gegevens geheim. Voor inzage door deze personen vragen wij u toestemming te geven. De Inspectie Gezondheidszorg en Jeugd kan zonder uw toestemming uw gegevens inzien.

We bewaren uw gegevens 15 jaar in het UMCG. Uw lichaamsmateriaal wordt maximaal voor dezelfde tijd in het UMCG bewaard. Het bewaren van uw gegevens en lichaamsmateriaal doen wij om daarop in de loop van het onderzoek nog nieuwe bepalingen te kunnen doen die te maken hebben met dit onderzoek. Uw lichaamsmateriaal wordt vernietigd zodra dit niet meer nodig is, de verzamelde gegevens worden wel bewaard.

Uw verzamelde gegevens en uw (overgebleven) lichaamsmateriaal kunnen ook van belang zijn voor ander wetenschappelijk onderzoek op het gebied van vitaliteit in melanoom patiënten. Daarvoor zullen uw gegevens en lichaamsmateriaal 15 jaar worden bewaard in het UMCG. In het toestemmingformulier geeft u aan of u dit goed vindt. Wanneer u dit niet wilt, kunt u nog steeds meedoen met dit onderzoek.

Om meer te weten te komen over uw rechten bij de verwerking van persoonsgegevens kunt u terecht op <u>www.autoriteitpersoonsgegevens.nl</u>. Wanneer u vragen heeft over uw rechten, neem dan contact op met degene die verantwoordelijk is voor de verwerking van uw persoonsgegevens. Voor uw onderzoek is dat het UMCG; zie **bijlage A** voor contactgegevens, en website.

Als u klachten heeft over de verwerking van uw persoonsgegevens, raden we u aan om deze eerst te bespreken met het onderzoeksteam. U kunt ook naar de Functionaris Gegevensbescherming van het UMCG gaan. Of u dient een klacht in bij de Autoriteit Persoonsgegevens.

Meer informatie over het onderzoek kunt u vinden op <u>www.ClinicalTrials.gov</u> Na het onderzoek kan de website een samenvatting van de resultaten van dit onderzoek tonen. U vindt het onderzoek door te zoeken op [TRIALCODE].

## 11. Vergoedingen

De onderzoeksmiddelen en testen die voor het onderzoek gebruikt worden kosten u niets. U krijgt ook geen vergoeding als u meedoet aan dit onderzoek. Wel krijgt u een vergoeding voor uw (extra) reiskosten. Deze kosten worden berekend op basis van 0.21 cent/km gereisd, reizen met 2° klas openbaar vervoer wordt ook volledig vergoed.

## 12. Verzekering

U bent niet extra verzekerd voor dit onderzoek. Want meedoen aan het onderzoek heeft geen extra risico's. Daarom hoeft de hoofdonderzoeker, gebaseerd op het besluit van de medisch-ethische toetsingscommissie, geen extra verzekering af te sluiten.

# 13. Vragen

Vragen over het onderzoek kunt u stellen aan de onderzoeker (E. Oosterhout, promovendus UMCG) of het hoofd van het onderzoek (Prof. Dr. G.A.P. Hospers, internist-oncoloog UMCG). Klachten kunt u bespreken met de onderzoeker of de arts die u behandelt. U kunt hiervoor ook terecht bij de Klachten Functionaris van het Universitair Medisch Centrum Groningen (UMCG). Voor spoedeisende gevallen kunt u bellen naar het algemene UMCG-nummer 050-3616161. Alle contactgegevens vindt u in **bijlage A**.

# 14. Toestemming voor deelname aan het onderzoek

U kunt eerst rustig nadenken over dit onderzoek. Daarna vertelt u de onderzoeker of u de informatie begrijpt en of u wel of niet wilt meedoen. Wanneer u besluit mee te willen doen aan het onderzoek vult u het toestemmingsformulier in dat u bij deze informatiebrief vindt. U en de onderzoeker krijgen allebei een getekende versie van deze toestemmingsverklaring.

Dank voor uw tijd.

E. Oosterhout, MSc Promovendus, UMCG
Prof. Dr. B.L. van Leeuwen Oncologisch chirurg, UMCG
Prof. Dr. G.A.P. Hospers Internist oncoloog, UMCG
Dr. R.J. Björk Postdoc onderzoeker, UMCG

Prof. Dr. R.K. Weersma MDL-arts, UMCG

# 15. Bijlagen

Bijlage A: Contact gegevens

Bijlage B: Overzicht afspraken en onderzoeken

Bijlage C: Ontlasting verzamelinstructie Bijlage D: Toestemmingsformulier

# Bijlage A: Contactgegevens voor Universitair Medisch Centrum Groningen

Hoofdonderzoeker UMCG: Prof. Dr. G.A.P, internist-oncoloog

Telefoonnummer: +31652724185

Email: g.a.p.hospers@umcg.nl

Onderzoeker UMCG: E. Oosterhout, PhD kandidaat

Telefoonnummer: +31652764949

Email: <u>e.oosterhout@umcg.nl</u>

Overige onderzoekers: Prof. Dr. B.L. van Leeuwen, Oncologisch chirurg

Dr. R.J. Björk, Postdoc onderzoeker

Prof. Dr. R.K. Weersma, Maag-darm-lever arts

Onafhankelijk arts: Dr. T.J.N. Hiltermann, long-oncoloog

Telefoonnummer: 050-3616161

#### Klachten:

Onafhankelijke klachtenfunctionaris via +31 (0)50 361 22 20 secretariaat, of <u>klachtenfunctionaris@umcg.nl</u> of wanneer u klachten heeft over de behandeling, kunt u contact opnemen met het team Patiëntinformatie via +31(0)50 361 3300 of <u>patientinformatie@bvl.umcg.nl</u>

Functionaris voor de Gegevensbescherming van de instelling:

Te bereiken: mevrouw B.M.Y. Sieperda, telefonisch +31(0)50 361 48 36 of secretariaat afd. Juridische zaken, +31(0)10 7034986 of <a href="mailto:privacy@umcg.nl">privacy@umcg.nl</a>

Voor meer informatie over uw rechten: op <u>uwprivacy.umcg.nl</u> of <u>www.autoriteitpersoonsgegevens.nl</u>

# Bijlage B: Overzicht afspraken en onderzoeken

Onderstaande tabel geeft een beknopt overzicht van de afspraken en onderzoeken aan. Voor een uitgebreide uitleg, zie dan de tekst onder de tabel. De schematische weergave van de tijdlijn van het onderzoek kunt u vinden in **figuur 1**.

| | Voor de<br>studie | Start van<br>studie<br>(T0) | Na 3<br>weken<br>(T1) | Na 6<br>weken<br>(T2) |
|---|---|---|---|---|
| Lezen van de studie informatie en tekenen toestemmingsformulier | Х | | | |
| Onderzoeksmiddel gebruiken | | Х | Х | Х |
| Bezoek aan ziekenhuis | | Х | Х | Х |
| Klinische evaluatie van eventuele bijwerkingen | | Х | Х | Х |
| Verzamelen van persoonsgegevens en gezondheidsgegevens | | Х | | |
| Lichaamsmetingen | | X | | |
| Bloed laten prikken in het ziekenhuis | | Х | Х | Х |
| Ontlasting opvangen thuis (1-3 dagen voor de onderzoek afspraak) en inleveren | | Х | Х | X |
| Voedselvragenlijst invullen | | Х | | X |
| Invullen van vragenlijsten, digitaal of op papier en meenemen of opsturen naar het ziekenhuis | | Х | Х | Х |

## Lezen van de informatiebrief en invullen van het toestemmingsformulier

Voor de studie ontvangt u deze informatiebrief en een toestemmingsformulier (**bijlage D**). U leest deze informatie rustig door en bedenkt of u mee wilt doen. Deze brief en het toestemmingsformulier neemt u mee naar uw vervolgafspraak. Na toestemming zal er contact met u opgenomen worden.

## Opnemen in de studie en het maken van de eerste onderzoek afspraak (30 minuten)

De onderzoeker zal met u telefonisch contact opnemen nadat u interesse heeft getoond om geïncludeerd te worden in de studie. U zult gevraagd worden over uw medische geschiedenis en het onderzoek zal nog kort besproken worden. Ten tweede, zal de onderzoeker uitleg geven over de vragenlijsten en het verzamelen van uw ontlasting, welke u beide voor de eerste onderzoek afspraak voldaan dient te hebben. Het is belangrijk dat u na dit gesprek het toestemmingsformulier getekend retourneert aan de onderzoeker. Aan het einde van het gesprek zal de eerste onderzoek afspraak zal er met u ingepland worden.

## Invullen van vragenlijsten (1 uur)

De onderzoeker zal u uitleg geven over de vragenlijsten die u digitaal of per post toegestuurd krijgt. U wordt verzocht vragenlijsten in te vullen over uw voedingspatroon, gesteldheid van de darmen en de kwaliteit van leven. Er wordt van u gevraagd om deze thuis in te vullen vóór het eerste bezoek. Deze vragenlijsten worden ook toegestuurd voor de volgende twee onderzoek afspraken, en er wordt van u gevraagd om deze vóór de afspraak thuis in te vullen.

## Verzamelen van ontlasting (10-20 minuten)

U verzamelt zelfstandig thuis uw ontlasting met behulp van het ontlasting verzamelpakket wat u ontvangt van de onderzoeker. Hoe u ontlasting verzameld vindt u in **bijlage C**. Het verzamelen van ontlasting kunt u 1-3 dagen voordat de afspraak met de onderzoeker plaatsvindt doen. U neemt de ontlasting mee naar de onderzoek afspraak in de koeltas die in het ontlasting verzamelpakket zit. Met het ontlasting onderzoek testen we de samenstelling van de bacteriën in uw darmen, aanwezigheid van korte-keten vetzuren en waardes die mate van ontsteking kunnen aantonen (calprotectine).

## Onderzoek afspraken (1 uur)

Tijdens het eerste bezoek zult u uitleg ontvangen over het onderzoeksmiddel en zal u uitgelegd worden hoe en wanneer u deze zal innemen. De zakjes met onderzoeksmiddel ontvangt u tijdens dit eerste bezoek.

Bij het eerste bezoek worden lichaamsmetingen uitgevoerd (gewicht, lengte, buikomtrek, bloeddruk). Verder zullen de ingevulde vragenlijsten ingenomen en gecontroleerd worden. Als laatste zal u gevraagd worden om bloed te laten afnemen, de onderzoeker zal u hiervoor naar de prikpoli verwijzen. Per keer wordt 1 buisje bloed afgenomen, wat gelijk staat aan 10 ml bloed. Het bloedonderzoek bestaat uit het isoleren van witte bloedcellen en plasma onderzoek.

## Schematische weergave van de onderzoeksperiode



# Bijlage C: Ontlasting verzamelinstructie

In deze instructie leest u welke materialen u van het onderzoeksteam ontvangt voor het verzamelen van ontlasting. In de beschrijving leest u stap voor stap hoe u de ontlasting thuis verzamelt. U wordt aangeraden de instructie eerst helemaal door te lezen voordat u daadwerkelijk de ontlasting gaat verzamelen.

Heeft u vragen over het verzamelen van ontlasting? Neem dan gerust contact met ons op.

U verzamelt de ontlasting thuis op één moment in de drie dagen voorafgaand aan de dag dat u een onderzoek afspraak heeft. Indien u bijvoorbeeld op woensdag een afspraak heeft; kunt u op zondag, maandag of dinsdag de ontlasting verzamelen. U vult alle buisjes in één keer.

Het opvangen en bewaren van de ontlasting verloopt in zes stappen.

- Opvangen van de ontlasting
- Verzamelen van ontlasting in de pipet
- Overbrengen van ontlasting in de pipet naar buisje
- Verzamelen van ontlasting met gebruik van een schepje
- Buisjes verzamelen in het zwarte zakje
- Bewaren van het zwarte zakje met de buisjes in de vriezer

In dit document worden de stappen nader toegelicht.

## Materialen

Om de ontlasting te kunnen verzamelen ontvangt u de volgende materialen (controleer uw ontlasting verzamelpakket):

- 1x Grijs opvangbakje
- 1x Handschoenen
- 1x Ontlasting opvanger
- 1x Schaar (alleen aanwezig in het eerste pakket)
- 3x Buisjes
- 1x Buisje met schepje
- 3x Plastic pipet
- 1x Zwart zakje
- 1x Doorzichtig zakje
- 1x Koeltas (alleen aanwezig in het eerste pakket)
- 1x Ontlastingsverzamelformulier

## Stap 1: Opvangen van de ontlasting

Om ontlasting op te vangen, gebruikt u de meegeleverde ontlasting opvanger.

- 1. Vouw voorzichtig de ontlasting opvanger open in de richting van de pijltjes.
- 2. Bevestig deze met de plakstroken op het achterste deel van de wc-bril, zonder dat de plakstrip met het water in contact komt.
- 3. Vang de ontlasting op.



## Stap 2: Verzamelen van ontlasting in de pipet

Na opvangen van de ontlasting, kunt u met de pipet de ontlasting verzamelen. Gebruik voor deze stap de handschoenen.

- 1. Knijp het ballonnetje bovenaan de pipet voorzichtig in en houd het uiteinde van de pipet in de ontlasting.
- 2. Druk de pipet tot ongeveer het eerste zwarte streepje in de ontlasting en laat het ballonnetje voorzichtig los. Door het loslaten van het ballonnetje kan de ontlasting een beetje omhoog gezogen worden, dat is niet erg.
- 3. Veeg de buitenkant van de pipet af met wc-papier.



## Stap 3: Overbrengen van ontlasting in de pipet naar buisje

Herhaal stap 2 en 3 zodat u in totaal 3 kleine buisjes met een pipet ontlasting heeft verzameld.

- 1. Breng het uiteinde van de pipet over in het kleine buisje met de schroefdop. Probeer hierbij geen contact te maken met de schroefdraad.
- 2. Knip het stukje pipet dat in het buisje zit af bij het tweede zwarte streepje.
- 3. Het stukje pipet wat overblijft kunt u weggooien in de prullenbak.







# Stap 4: Verzamelen ontlasting met gebruik van een schepje

- Draai de dop met het schepje van de buis af.
- Steek het schepje in de ontlasting.
- Schep de ontlasting op.
- Breng het schepje naar het buisje en vul het buisje maximaal tot de helft. Probeer hierbij geen contact te maken met het schroefdraad van het buisje.



## Stap 5: Buisjes verzamelen in het zwarte zakje

- 1. Doe de drie kleine buisjes en het buisje met schepje rechtop in het zwarte zakje.
- 2. Vul het ontlastingsverzamelingsformulier in en steek deze ook in het zwarte zakje.
- 3. Doe het zwarte zakje in het doorzichtige zakje, zorg ervoor dat uw gegevens zichtbaar blijven.

## Stap 6: Bewaar het zwarte zakje met de buisjes in de vriezer

- 1. Plaats de verzamelde materialen direct in de vriezer.
- 2. Bewaar het zwarte zakje in de vriezer tot de onderzoek afspraak, u neemt het zwarte zakje in de koeltas mee naar de afspraak.

Het verzamelen van ontlasting is nu klaar en de ontlasting opvanger kan nu doorgespoeld worden. Wacht voor het doorspoelen een ogenblik, zodat het papier wat water opneemt en makkelijker door te spoelen is. Het grijze bakje kan in de afvalbak of container.

# Bijlage D: Toestemmingsformulier deelnemer

# ONDERZOEK NAAR DE EFFECTEN VAN VEZELRIJKE GEDROOGDE WITLOFWORTEL OP HET DARM MICROBIOOM BIJ OPERATIEF BEHANDELDE MELANOOM PATIËNTEN

- Ik heb de informatiebrief gelezen. Ook kon ik vragen stellen. Mijn vragen zijn goed genoeg beantwoord.
- Ik had genoeg tijd om te beslissen of ik meedoe.
- Ik weet dat meedoen vrijwillig is. Ook weet ik dat ik op ieder moment kan beslissen om toch niet mee te doen met het onderzoek. Of om ermee te stoppen. Ik hoef dan niet te zeggen waarom ik wil stoppen.
- Ik geef de onderzoeker toestemming om mijn huisarts, behandelend specialist en apotheker te laten weten dat ik meedoe aan dit onderzoek.
- Ik geef de onderzoeker toestemming om informatie op te vragen bij mijn huisarts en/of de specialist die mij behandelt over mijn ziektegeschiedenis en medicatiegebruik.
- Ik geef de onderzoeker toestemming om mijn huisarts of specialist informatie te geven over onverwachte bevindingen uit het onderzoek die van belang zijn voor mijn gezondheid.
- Ik geef de onderzoekers toestemming om mijn gegevens en lichaamsmateriaal te verzamelen en gebruiken.
   De onderzoekers doen dit alleen om de onderzoeksvraag van dit onderzoek te beantwoorden en om het middel te laten registreren.
- Ik weet dat voor de controle van het onderzoek sommige mensen al mijn gegevens kunnen inzien. Die mensen staan in deze informatiebrief. Ik geef deze mensen toestemming om mijn gegevens in te zien voor deze controle.
- Ik wil meedoen aan dit onderzoek.

Wilt u in de tabel hieronder ja of nee aankruisen?

| Ik geef toestemming om mijn gegevens te bewaren om dit te gebruiken voor ander onderzoek, zoals in de informatiebrief staat. | Ja □ | Nee □ |
|---|---|---|
| Ik geeft toestemming om mijn (overgebleven) lichaamsmateriaal te bewaren om dit te | | Nee □ |
| gebruiken voor ander onderzoek, zoals in de informatiebrief staat. Het lichaamsmateriaal | | |
| wordt daarvoor nog 15 jaar bewaard. | | |
| Ik geef toestemming om mij eventueel na dit onderzoek te vragen of ik wil meedoen met | | Nee □ |
| een vervolgonderzoek. | | |
| Ik geef de onderzoekers toestemming om na het onderzoek de belangrijkste uitkomsten | | Nee □ |
| met mij te delen. | | |

| Naam (proefpersoon): | |
|---|---|
| Handtekening: | Datum: / / |
| | nformeerd over het genoemde onderzoek. Wanneer er |
| | e toestemming van de proefpersoon kan beïnvloeden, |
| dan laat ik dit op tijd weten aan deze proefpersoon. | |
| Naam (onderzoeker of vertegenwoordiger): | |
| Handtekening: | <br>Datum: / / |
| Aanvullende informatie is gegeven door: | |
| Administrate in Septem about | |
| Naam: | |
| Functie: | |
| Handtekening: | Datum: / / |
| | matiebrief mee, samen met de getekende versie van het |
| toestemmingsformulier. | |